CLINICAL TRIAL: NCT07211451
Title: Low Axillary Nodal Metastasis Rates in Selected HER2-Positive and Triple-Negative Breast Cancer Patients: Toward De-escalation of Sentinel Lymph Node Biopsy
Brief Title: Axillary Nodal Burden in HER2+ and TNBC
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professpr, Gangnam Severance Hospital
Other Study IDs: 3-2025-0126
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Sentinel lymph node biopsy; Omission; HER2; Triple-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Breast conserving surgery with axillary surgery — In this study, all patients received breast conserving surgery with axillary surgery.

SUMMARY:
This study aimed to evaluated rates of pathologic axillary nodal metastasis in patients with with early-stage HER2-positive BC or TNBC who had clinically node-negative status on preoperative ultrasonography and underwent upfront breast-conserving surgery (BCS) with axillary surgery. In addition, this study aimed to identify subgroups in which SLNB omission may be feasible.

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive breast cancer or TNBC
* Patients who received upfront breast conserving surgery with axillary surgery
* Patients who had a clinically axillary node negative disease

Exclusion Criteria:

* Patients who underwent mastectomy
* Absence of axillary nodal assessment on ultrasonography
* Patients who underwent mastectomy
* Patients who underwent mastectomy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early-stage HER2-positive breast cancer or TNBC who had clinically node-negative status on preoperative ultrasonography and underwent upfront breast-conserving surgery (BCS) with axillary surgery
Sampling Method: Non-Probability Sample
Enrollment: 1571 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Pathologic axillary lymph node metastasis rate | Immediately after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, Please Select, South Korea

IPD SHARING:
Plan to Share IPD: No